CLINICAL TRIAL: NCT03171610
Title: Randomized Double-blind Study on Efficacy of iv PCA With Fentanyl or Sufentanil in Patients Undergoing Laparoscopic Nephrectomy
Brief Title: Study on Efficacy of iv PCA With Fentanyl or Sufentanil in Patients Undergoing Laparoscopic Nephrectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 4-2017-0201
Record Dates: First submitted 2017-05-22; First posted 2017-05-31 (Actual); Last update posted 2018-03-15 (Actual); Status verified 2018-03

CONDITIONS: Patients Undergoing Laparoscopic Nephrectomy
Keywords: laparoscopic nephrectomy; Patient-controlled analgesia (PCA); sufentanil; fentanyl

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sufentanil group (Experimental): Arm Description: PCA with sufentanil (3 mcg/kg), ramosetron (NaseaTM) 0.3 mg and ketorolac 120 mg in a normal saline with a total volume of 100ml
  Interventions: Drug: Sufentanil group
- Fentanyl group (Active Comparator): PCA with fentanyl (20 mcg/kg), ramosetron (NaseaTM) 0.3 mg and ketorolac 120 mg in a normal saline with a total volume of 100ml
  Interventions: Drug: Fentanyl group

INTERVENTIONS:
Drug: Sufentanil group — PCA device containing sufentanil (3 mcg/kg), ramosetron (NaseaTM) 0.3 mg and ketorolac 120 mg in a normal saline with a total volume of 100ml was connected.
  Arms: Sufentanil group
Drug: Fentanyl group — PCA device containing fentanyl (20 mcg/kg), ramosetron (NaseaTM) 0.3 mg and ketorolac 120 mg in a normal saline with a total volume of 100ml was connected.
  Arms: Fentanyl group

SUMMARY:
The purpose of this study is to compare the efficacy of iv PCA with fentanyl or sufentanil in patients undergoing laparoscopic nephrectomy

ELIGIBILITY:
Inclusion Criteria:

1. patients undergoing laparoscopic or robot-assisted laparoscopic nephrectomy (total or partial)
2. patient who want intravenous PCA for postoperative pain control

Exclusion Criteria:

1. long-term use of opioid, pain reliever or tranquilizers
2. a history of DM neuritis
3. prolonged prothrombin time or activated partial thromboplastin time
4. impairment of cognitive function
5. obesity (BMI ≥ BMI 30 kg/m2)

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2017-06-13 (Actual); Primary Completion 2018-01-03 (Actual); Study Completion 2018-01-03 (Actual)

PRIMARY OUTCOMES:
Efficacy of iv PCA with fentanyl or sufentanil in patients undergoing laparoscopic nephrectomy: Incidence of postoperative nausea and vomiting (PONV) | 24 hrs after recovery room discharge
  Incidence of postoperative nausea and vomiting (PONV)

SECONDARY OUTCOMES:
postoperative pain score | at arrival to recovery room, 30 minutes after arrival to recovery room, 1 hour after recovery room discharge, 6 hrs after recovery room discharge, 24 hrs after recovery room discharge
  NRPS (numerical verbal rating score of pain)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Yonsei University College of Medicine, Seoul, Korea, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No